CLINICAL TRIAL: NCT05093322
Title: An Open-Label, Multicenter Phase 1/2 Study of Surufatinib in Combination With Gemcitabine in Pediatric, Adolescent, and Young Adult Patients With Recurrent or Refractory Solid Tumors
Brief Title: A Study of Surufatinib in Combination With Gemcitabine in Pediatric, Adolescent, and Young Adult Patients With Recurrent or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2020-012-GLOB2; 2021-003602-41 (EudraCT Number)
Expanded Access: NCT04814732 (No longer available)
Record Dates: First submitted 2021-09-20; First posted 2021-10-26 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: Solid Tumor; Lymphoma; Osteosarcoma; Ewing Sarcoma; Rhabdomyosarcoma; Non-rhabdomyosarcoma Soft Tissue Sarcoma (NRSTS)
MeSH Terms: conditions — Lymphoma; Osteosarcoma; Sarcoma, Ewing; Rhabdomyosarcoma; Sarcoma | interventions — surufatinib; Gemcitabine

STUDY DESIGN:
Intervention Model Description: The study will be conducted in 2 parts:
  Part 1 - evaluation of tolerability and safety of surufatinib administered in combination with gemcitabine, and confirmation of the recommended clinical dose of surufatinib in pediatric patients with recurrent or refractory solid tumors or lymphoma. Part 2 - evaluation of anti-tumor activity and confirmation of tolerability of surufatinib administered in combination with gemcitabine in pediatric patients with recurrent or refractory osteosarcoma, Ewing sarcoma, RMS, and NRSTS.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1- Dose escalation (Experimental): Dose escalation study with sequential dose escalation of surufatinib in combination with gemcitabine. Patients with any recurrent or refractory solid tumors or lymphoma, who have a known or expected dysfunction of VEGFR-1, -2, and -3; FGFR-1; or CSF-1R pathways may be enrolled.
  Interventions: Drug: Surufatinib in combination with Gemcitabine
- Part 2 - Dose expansion (Experimental): Once the MTD/RP2D has been determined in the part 1 portion of the study, the part 2 disease specific cohorts for patients with refractory or recurrent osteosarcoma, Ewing Sarcoma, and RMS and NRSTS will open for enrollment.
  Interventions: Drug: Surufatinib in combination with Gemcitabine

INTERVENTIONS:
Drug: Surufatinib in combination with Gemcitabine — Surufatinib in combination with Gemcitabine
  Other Names: HMPL-012, sulfatinib in combination with Gemcitabine

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of surufatinib, thereby identifying the Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) of surufatinib administered in combination with gemcitabine in pediatric patients with recurrent or refractory solid tumors or lymphoma. The study will be conducted in 2 parts.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and tolerability of surufatinib, thereby identifying the Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) of surufatinib administered in combination with gemcitabine in pediatric patients with recurrent or refractory solid tumors or lymphoma. The study will be conducted in 2 parts:

Part 1 - evaluation of tolerability and safety of surufatinib administered in combination with gemcitabine, and confirmation of the recommended clinical dose of surufatinib in pediatric patients with recurrent or refractory solid tumors or lymphoma.

Part 2 - evaluation of anti-tumor activity and confirmation of tolerability of surufatinib administered in combination with gemcitabine in pediatric patients with recurrent or refractory osteosarcoma, Ewing sarcoma, RMS, and non-rhabdomyosarcoma soft tissue sarcoma (NRSTS).

Part 1 will enroll 2 to 6 patients per dose level cohort (up to 4 cohorts) with recurrent or refractory solid tumors. During cycle 1, surufatinib will be administered, orally, once daily (QD), as a single agent for 14 days followed by surufatinib daily in combination with gemcitabine intravenously on days 15 and 22 (cycle 1 duration=35 days) and days 1 and 8 of all subsequent cycles (cycle duration=21 days). Assessment based on dose limiting toxicity (DLT) criteria will be performed in the first 35-day cycle (DLT Evaluation Period). This study will utilize a rolling 6 design for part 1, with 3 dose escalation levels and 1 de escalation level, if needed.

Part 2 of the study will use a Simon 2-stage design with a maximum of 18 patients per cohort (osteosarcoma, Ewing sarcoma, RMS, and non-rhabdomyosarcoma soft tissue sarcoma (NRSTS)).

Surufatinib will be administered orally at identified MTD/RP2D daily in combination with gemcitabine (1000 mg/m2 weekly × 2 doses) intravenously on days 1 and 8.

In both parts 1 and 2, patients can remain on treatment until completing cycle 17, or until progressive disease, unacceptable toxicity, or death; whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Age: At time of study enrollment, patients must be

   For US Sites:
   1. Part 1 (including PK expansion cohort): ≥2 and <18 years of age;
   2. Part 2: ≥2 and ≤18 years of age;

   For EU/UK Sites:
   1. Part 1 (including PK expansion cohort): from birth to <18 years of age;
   2. Part 2: from birth to <18 years of age (except as noted below);

      * Note: Patients <2 years of age will only be enrolled in Europe, however, enrollment of patients <2 years of age will not begin until definitive juvenile animal toxicity data is available.
2. Diagnosis:

   1. Part 1 - Patients with any recurrent or refractory solid tumors or lymphoma (not central nervous system [CNS]) that have a known or expected dysfunction of VEGFR 1, -2, and -3; FGFR-1, or CSF-1R pathways (based on literature) are eligible. Patients must have had histologic verification of malignancy at original diagnosis or relapse.
   2. Part 2 - Recurrent or refractory osteosarcoma (US and EU), Ewing sarcoma (US and EU), RMS (US and EU), or NRSTS (EU only). Patients must have had histologic verification of malignancy at original diagnosis or relapse.
3. Disease status: Patients must have measureable or evaluable disease for part 1 dose escalation; for part 2, patients must have measurable disease by RECIST version 1.1.
4. Therapeutic options: Patient's current disease state must be one for which there is no known curative therapy.
5. Performance level: Karnofsky ≥50 for patients ≥16 and <18 years of age and Lansky ≥50 for patients <16 years of age, Eastern Cooperative Oncology Group (ECOG) ≤2 for patients ≥18 years of age.
6. Adequate organ and bone marrow function as defined in the current protocol.
7. Adequate cardiac function as indicated as defined in the current protocol.
8. Patients with known bone marrow metastatic disease will be eligible for the study provided they meet the blood counts in the inclusion criteria as defined in the current protocol.
9. Adequate BP control which is defined as a BP <95th percentile (≤ grade 1) for age, height, and sex.
10. Informed consent: Provision of signed and dated written informed consent (parent/legal guardian if patient <18 years of age) and assent (from patients aged >7 years) prior to any study-specific procedures, sampling, and analyses.
11. Patient must meet all defined Inclusion criteria as defined in the current protocol.

Exclusion Criteria:

1. Patient must not meet any exclusion criteria as defined in the current protocol.
2. Pregnant, breast feeding or planning on becoming pregnant.
3. Patients is taking and prohibitive concomitant medications as outlined in the current protocol.
4. Patients have an uncontrolled infection.
5. Patients has had major surgery or significant traumatic injury within 28 days of the first dose.
6. Brain metastases and/or spinal cord compression untreated with surgery and/or radiotherapy and without clinical imaging evidence of SD for 14 days or longer.
7. History of allergies to Surufatinib and/or Gemcitabine.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josephine Haduong, Principal Investigator — Children's Hospital of Orange County
Locations (11):
- United States (11):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Childrens Hospital Orange County, Orange, California
  - Children's National Hospital, Washington D.C., District of Columbia
  - Riley Hospital for Children, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Seattle Children's Hospital, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 1/2 open-label study was conducted in pediatric, adolescent, and young adult patients with recurrent or refractory solid tumors at 8 study sites.
Pre-assignment Details: This study consisted of a screening period (up to 28 days), followed by a treatment phase (Cycle 1: 35 days and subsequent cycles: 21 days) and safety follow-up period (up to 30 days). A total of 13 patients were enrolled in this study. The planned expansion phase for this study was not opened.
Groups:
- Dose Level 1: Patients received surufatinib 120 milligram/meter square (mg/m^2) oral capsule once daily (QD) as a single agent for 14 days followed by surufatinib daily in combination with gemcitabine 1000 mg/m^2/dose intravenous (IV) infusion on Days 15 and 22 of a 35-day Cycle 1 and on Days 1 and 8 of 21-day subsequent cycles until progressive disease (PD), unacceptable toxicity, or death; whichever came first.
- Dose Level 2: Patients received surufatinib 160 mg/m^2 oral capsule QD as a single agent for 14 days followed by surufatinib daily in combination with gemcitabine 1000 mg/m^2/dose IV infusion on Days 15 and 22 of a 35-day Cycle 1 and on Days 1 and 8 of 21-day subsequent cycles until PD, unacceptable toxicity, or death; whichever came first.
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2
Started | 10 | 3
Completed | 0 | 0
Not Completed | 10 | 3
Not completed — Death | 6 | 2
Not completed — Other | 4 | 1

BASELINE CHARACTERISTICS:
Population: The Safety analysis set included all patients who received at least 1 dose of surufatinib or gemcitabine.
Groups:
- Dose Level 1: Patients received surufatinib 120 mg/m^2 oral capsule QD as a single agent for 14 days followed by surufatinib daily in combination with gemcitabine 1000 mg/m^2/dose IV infusion on Days 15 and 22 of a 35-day Cycle 1 and on Days 1 and 8 of 21-day subsequent cycles until PD, unacceptable toxicity, or death; whichever came first.
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Total
Number analyzed (Participants) | 10 | 3 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.8 (5.55) | 13.7 (2.89) | 12.2 (5.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 6 | 2 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 9 | 1 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2 | 0 | 2
  White | 7 | 2 | 9
  Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose-Limiting Toxicities (DLT)
Description: A DLT was defined as any of following events that were attributable to study treatment (at least possibly related). Adverse events (AE) were graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
  * Any Grade 3 or greater nonhematological toxicity.
  * Grade 3 liver enzyme elevation.
  * Cases of Hy's law.
  * Any Grade 2 nonhematological toxicity that persisted for >= 7 days.
  * Any Grade 4 hypertension.
  * Grade 3 corrected QT interval prolongation > 500 millisecond.
  * Grade 4 thrombocytopenia for > 7 days.
  * Grade 3 thrombocytopenia with clinically significant bleeding.
  * Grade 4 neutropenia that lasted for > 7 days.
  * Myelosuppression that caused a delay of > 7 days in the start of Cycle 2.
Time Frame: From the first dose of study drug (Day 1) up to Day 35 of Cycle 1
Population: The DLT evaluable set included all patients enrolled in dose escalation phase of study who received at least 80% of surufatinib dose and both doses of gemcitabine during DLT evaluation period or who discontinued treatment due to a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 8 | 3
Participants | 0 | 2

2. Primary Outcome: Number of Patients With Treatment Emergent Adverse Events (TEAEs) by Severity
Description: The AEs were graded using the NCI CTCAE version 5.0. The CTCAE displays Grades 1 through 5 where, Grade 1= mild, Grade 2= moderate, Grade 3= Severe, Grade 4= life-threatening consequences and Grade 5= death.
Time Frame: From the first dose of study drug (Day 1) up to 30 + 7 days after the last dose of study drug, approximately 19 weeks
Population: The Safety analysis set included all patients who received at least 1 dose of surufatinib or gemcitabine.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 10 | 3
Participants
  Grade 1 | 0 | 0
  Grade 2 | 1 | 1
  Grade 3 | 4 | 2
  Grade 4 | 3 | 0
  Grade 5 | 2 | 0

3. Primary Outcome: Number of Patients With Clinically Significant Physical Examination Abnormalities
Description: Physical examination included patient height, weight, and general condition, as well as an examination of the head, heart, chest (including the lungs), abdomen, extremities, skin, lymph nodes, nervous system, and additional areas/systems as clinically indicated.
Time Frame: From the first dose of study drug (Day 1) up to 30 + 7 days after the last dose of study drug, approximately 19 weeks
Population: The Safety analysis set included all patients who received at least 1 dose of surufatinib or gemcitabine.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 10 | 3
Participants | 6 | 1

4. Primary Outcome: Number of Patients With Clinically Significant Vital Signs Abnormalities
Description: Vital signs included systolic blood pressure (BP), diastolic BP, heart rate, height, weight, respiratory rate, and body temperature.
Time Frame: From the first dose of study drug (Day 1) up to 30 + 7 days after the last dose of study drug, approximately 19 weeks
Population: The Safety analysis set included all patients who received at least 1 dose of surufatinib or gemcitabine.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 10 | 3
Participants | 0 | 0

5. Primary Outcome: Number of Patients With Clinically Significant Laboratory Abnormalities
Description: Blood and urine samples were collected to determine the clinical chemistry, hematology, and urinalysis laboratory abnormalities.
Time Frame: From the first dose of study drug (Day 1) up to 30 + 7 days after the last dose of study drug, approximately 19 weeks
Population: The Safety analysis set included all patients who received at least 1 dose of surufatinib or gemcitabine.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 10 | 3
Participants | 0 | 1

6. Primary Outcome: Number of Patients With Clinically Significant 12-Lead Electrocardiogram (ECG) Abnormalities
Description: Standard 12-lead ECGs were performed after the patient rested for 5 to 10 minutes. The ECG parameters included heart rate, PR interval, RR interval, QT interval, QTcF, and QRS interval from the triplicate 12-lead ECG.
Time Frame: From the first dose of study drug (Day 1) up to 30 + 7 days after the last dose of study drug, approximately 19 weeks
Population: The Safety analysis set included all patients who received at least 1 dose of surufatinib or gemcitabine.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 10 | 3
Participants | 1 | 0

7. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR was defined as the percentage of patients with a best overall response (BOR) of complete response (CR) or partial response (PR) as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. The BOR was defined as the best response recorded from the start of study treatment until documented RECIST version 1.1 progression, death, or withdrawal of consent. The CR was defined as disappearance of all target lesions. The PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: RECIST assessments performed at baseline (within 28 days before start of study treatment), Day 1 of Cycle 3 and until confirmed objective disease progression. Up to approximately 19 weeks.
Population: The Safety analysis set included all patients who received at least 1 dose of surufatinib or gemcitabine.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 10 | 3
percentage of patients | 0 [0.0 to 30.8] | 0 [0.0 to 70.8]

8. Secondary Outcome: Disease Control Rate (DCR)
Description: The DCR was defined as the percentage of patients with a BOR of CR, PR, or stable disease as determined by the investigator using RECIST version 1.1. Stable disease was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum on study.
Time Frame: as for outcome 7
Population: The Safety analysis set included all patients who received at least 1 dose of surufatinib or gemcitabine.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 10 | 3
percentage of patients | 20.0 [2.5 to 55.6] | 0 [0.0 to 70.8]

9. Secondary Outcome: Time to Response (TTR)
Description: The TTR was defined as the time from the start of study treatment until the date of the first occurrence of PR or CR for responders only.
Time Frame: as for outcome 7
Population: The Safety analysis set included all patients who received at least 1 dose of surufatinib or gemcitabine. No responders in this study.
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Duration of Response (DoR)
Description: The DoR was defined as the time from the first occurrence of PR or CR whichever came first, until disease progression or death.
Time Frame: as for outcome 7
Population: as for outcome 9
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Progression-Free Survival (PFS)
Description: The PFS was defined as the time from the start of study treatment until the first radiographic documentation of objective progression as assessed by the investigator using RECIST version 1.1 or death from any cause.
Time Frame: as for outcome 7
Population: The Safety analysis set included all patients who received at least 1 dose of surufatinib or gemcitabine.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 10 | 3
months | 1.8 [0.7 to NA] — The upper limit of 95% confidence interval could not be estimated either due to insufficient number of PFS events or not sufficient follow-up time at the time of the analysis. | 1.5 [1.1 to NA] — The upper limit of 95% confidence interval could not be estimated either due to insufficient number of PFS events or not sufficient follow-up time at the time of the analysis.

12. Secondary Outcome: Number of Patients Who Performed Taste and Palatability Survey of Surufatinib
Description: The taste and palatability survey was assessed in patients who had taken surufatinib oral suspension. For pediatric patients, their parents completed the taste and palatability survey. Data for the evaluation of taste of surufatinib oral suspension was summarized on a scale of 1 (very bad) through 5 (very nice).
Time Frame: Days 1 and 8 of Cycle 1
Population: The Safety analysis set included all patients who received at least 1 dose of surufatinib or gemcitabine. Only patients who performed the survey are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 2 | 0
Participants
  Cycle 1 Day 1: Very Nice | 0 |
  Cycle 1 Day 1: Nice | 1 |
  Cycle 1 Day 1: Not Nice, not Bad | 0 |
  Cycle 1 Day 1: Bad | 1 |
  Cycle 1 Day 1: Very Bad | 0 |
  Cycle 1 Day 8: Very Nice | 0 |
  Cycle 1 Day 8: Nice | 1 |
  Cycle 1 Day 8: Not Nice, not Bad | 0 |
  Cycle 1 Day 8: Bad | 1 |
  Cycle 1 Day 8: Very Bad | 0 |

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs (TEAEs) were collected from the first dose of study drug (Day 1) up to 30 + 7 days after the last dose of study drug, approximately 19 weeks
Description: The Safety analysis set included all patients who received at least 1 dose of surufatinib or gemcitabine.
Arm/Group | Dose Level 1 | Dose Level 2
All-Cause Mortality (participants affected / at risk) | 6/10 | 2/3
Serious Adverse Events (participants affected / at risk) | 7/10 | 1/3
Other Adverse Events (participants affected / at risk) | 10/10 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=10) | Dose Level 2 (N=3)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Disease progression (General disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Device breakage (Product Issues) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=10) | Dose Level 2 (N=3)
Hypertension (Vascular disorders) | 2 (3) | 2 (3)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (6) | 2 (2)
Fatigue (General disorders) | 3 (4) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (3) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 3 (5)
Neutrophil count decreased (Investigations) | 5 (9) | 1 (1)
Platelet count decreased (Investigations) | 4 (11) | 1 (1)
White blood cell count decreased (Investigations) | 3 (6) | 2 (3)
Activated partial thromboplastin time prolonged (Investigations) | 2 (4) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1)
International normalised ratio increased (Investigations) | 3 (5) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (7) | 1 (4)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (2) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 1 (2)
Blood bicarbonate decreased (Investigations) | 1 (2) | 0 (0)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (4) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 6 (16) | 2 (5)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 2 (4)
Leukopenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (5) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (10) | 2 (3)
Vomiting (Gastrointestinal disorders) | 5 (6) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (8) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (5) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 4 (6) | 1 (3)
Haematuria (Renal and urinary disorders) | 1 (2) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 2 (3) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (5) | 2 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (7) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (11) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (5) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT05093322/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT05093322/SAP_001.pdf